CLINICAL TRIAL: NCT06230666
Title: Single-isocenter SBRT vs. Multiple-isocenter SBRT for Multiple Extracranial Metastases: a Randomized Controlled Non-inferiority Clinical Trial
Brief Title: Single-isocenter SBRT vs. Multiple-isocenter SBRT for Multiple Extracranial Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matthias Guckenberger (Other)
Responsible Party: Sponsor-Investigator, Matthias Guckenberger, Professor, Dr., Chairman, Radiation Oncology Department, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-01904
Record Dates: First submitted 2023-12-05; First posted 2024-01-30 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-isocenter SBRT (Experimental): SBRT using a single-isocenter treatment plan
  Interventions: Radiation: SBRT
- Multiple-isocenter SBRT (Active Comparator): SBRT using multiple treatment plans
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Stereotactic Body Radiation Therapy

SUMMARY:
The goal of this randomized non-inferiority clinical trial is to investigate whether single-isocenter SBRT using one treatment plan is similarly effective as multiple-isocenter SBRT using multiple treatment plans for multiple extracranial metastases. The main question it aims to answer is:

- whether 1-year freedom from local disease progression at the site of treated metastases after single-isocenter SBRT is non-inferior against multiple-isocenter SBRT at the same prescription doses.

Cancer patients with multiple extracranial distant metastases will be randomly assigned and treated either with single-isocenter SBRT or multiple-isocenter SBRT.

DETAILED DESCRIPTION:
Treatment planning of SBRT for multiple metastases usually employs multiple isocenters, one for each target, resulting in multiple treatment plans. Execution of such treatments requires sequential multiple setups and treatment plan verifications. This practice complicates the workflow of SBRT planning and delivery and makes target-by-target treatment lengthy and patient compliance and comfort suboptimal. The investigators hypothesized that single-isocenter SBRT for extracranial multiple metastases is non-inferior in terms of local efficacy as compared to multiple-isocenter SBRT at the same radiation dose prescription.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH/GCP regulations signed and dated by the participant and the investigator before any trial specific procedures (Informed Consent Form);
* Distant extracranial metastases (lung, mediastinal/cervical lymph node, liver, bone including spinal/paraspinal and abdominal/pelvic) from histologically confirmed cancer;
* Distant metastases confirmed by imaging:

  * CT is required in all cases;
  * MRI is required for spinal and recommended for liver metastases;
  * PET/CT is recommended for tumors showing high uptake of 18F-FDG, 11Ccholine, 68Ga- or 18F-PSMA;
* At least 2 distant metastases that are amendable to treat with a single isocenter approach according to the judgment of the treating clinician;
* Patients who are willing and able to comply with scheduled visits, treatment, and other trial procedures.

Exclusion Criteria:

* Prior radiotherapy for distant metastases if overlapping previous and current treatment plans leads to excessive dose to OARs;
* Distant metastases with extension into the gastrointestinal tract, skin;
* Large inter-lesion distance and location of distant metastases in different organs with different motion patterns;
* Women who are pregnant or breast feeding;
* Intention to become pregnant during the course of the trial;
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases;
* Known or suspected non-compliance, drug or alcohol abuse;
* Inability to follow the procedures of the trial, e.g. due to language problems of the participant;
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Female participants who underwent hysterectomy and/or bilateral oophorectomy or postmenopausal for longer than 2 years are not considered as being of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from local disease progression at the site of treated metastases | 1 year post-SBRT
  Local control at the site of treated metastases

SECONDARY OUTCOMES:
Acute adverse events (AEs) | 3 months post-SBRT
  AEs occurring during SBRT and within 3 months post-SBRT
Late adverse events (AEs) | 12 months post-SBRT
  AEs occurring 3 months post-SBRT and later
Overall survival | 1 year post-SBRT
  The time from randomization to death from any cause
Progression-free survival | 1 year post-SBRT
  The time from randomization to cancer progression at any site or death, whichever comes first
Overall treatment time | During the procedure
  Time needed for setup, verification and beam-on

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Upon an individual request